CLINICAL TRIAL: NCT06251466
Title: A Monocenter, Randomized Controlled, Pilot Study of Telemonitoring for Gestational Diabetes Mellitus.
Brief Title: Telemonitoring of Pregnancies Complicated With Gestational Diabetes Mellitus.
Acronym: TEGEDIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dr. Dorien Lanssens, Doctor - navorser, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Z-2022147
Record Dates: First submitted 2024-01-09; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Gestational Diabetes; Telemonitoring
Keywords: Gestational outcomes; User-experience
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Participants are randomized in either the control group or the telemonitoring group. The control group receives the standard care of gestational diabetes mellitus, meaning that the participants need to call their blood glucose levels weekly to the endocrinology department. The telemonitoring group receives telemonitoring, meaning that the participants need to register their blood glucose levels weekly in a smartphone application which is coupled to a platform in the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring group (Experimental): Participants randomized in the telemonitoring group receive a glucose meter to monitor their blood glucose levels at home. They need to perform the same measurements as the control group. The only difference lies in how they transmit their blood glucose measurement to the hospital. After each measurement, they need to register these levels once a week in the iHealth Gluco-Smart application. This data is send, via Bluetooth and Wi-Fi, to an online dashboard, called Dharma, for review by the researchers of the Mobile Health Unit of Hospital Oost-Limburg (ZOL) in Genk. Participants measuring abnormal blood glucose levels at one of the four time points are requested to measure their blood glucose levels again on the following day. The researcher contacts the endocrinology department if any abnormal blood glucose values are detected. Interventions including, starting insulin treatment, will be performed by the endocrinologist when necessary.
  Interventions: Device: iHealth Gluco-Smart application
- Control group (No Intervention): Pregnant women randomized in the control group receive a glucose meter to monitor their blood glucose levels at home. They need to measure their blood glucose levels four times a week, including: before breakfast, two hours after breakfast, two hours after lunch, two hours after dinner. These values are then called by the pregnant women to the endocrinology department. Interventions including, starting insulin treatment, will be performed by the endocrinologist when necessary.

INTERVENTIONS:
Device: iHealth Gluco-Smart application — iHealth Gluco-Smart is an application where blood glucose measurements can be registered. This application can be coupled to a platform in the hospital, called Dharma, that enables the researchers to evaluate these blood glucose levels.
  Arms: Telemonitoring group

SUMMARY:
This interventional study examines the addition of telemonitoring (TM) in prenatal care for gestational diabetes mellitus (GDM). By incorporating TM into the prenatal care for GDM, it is expected to achieve faster and improved follow-up, resulting in faster reaction time in the detection of aberrant blood glucose levels. Therefore, the overarching aim is to improve maternal and newborn pregnancy outcomes through optimized monitoring strategies (TM).

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is characterized by the onset of spontaneous hyperglycemia, typically diagnosed in the second or third trimester of gestation. GDM can have short-term complications for both the mother and the unborn child, including neonates with macrosomia which can complicate delivery, necessitating a cesarean section. While GDM usually resolves following delivery, it can also have long-term consequences, including neonatal hypoglycemia, increased risk of developing maternal hypertension, and type 2 diabetes. Therefore, a proper follow-up, including monitoring of blood glucose values, plays a crucial role in preventing both the pregnant woman and the unborn child from potential complications.

The principal measures for blood glucose level regulation in GDM involve lifestyle modifications, comprising dietary adjustments and exercise, supplemented as necessary by intermittent insulin therapy. Together with these lifestyle modifications and/or insulin therapy, these pregnant women also need to measure their blood glucose values once a week at home at four different time points, including: before breakfast, two hours after breakfast, two hours after lunch, and two hours after dinner. These measurements are performed with a glucose meter and are called to the nurse of the endocrinology department. This medical information allows the endocrinologist to make treatment adjustments (low sugar diet or insulin therapy) when necessary, potentially preventing the need for hospitalization due to GDM-associated complications.

However, a limitation of this standard care lies in the potential oversight by pregnant women in monitoring and reporting their blood glucose values to the endocrinology department. Unfortunately, this may result in the delayed detection of alarming values. Additionally, it imposes an increased workload on nurses, as they are required to contact these patients on each occasion. Altogether, there is less effective follow-up, leading to an increased risk of developing GDM-complications for both the mother and neonate. This less effective follow-up may contribute to increased healthcare costs, particularly in situations where hospitalization is required due to GDM-related complications.

Adding telemonitoring (TM) to the standard care of pregnant women with GDM offers a viable solution to mitigate the limitation described above. TM can be defined as the use of telecommunication technologies to assist the transmission of medical information between the patient and the caregiver. Regarding the care of GDM, the pregnant women are expected to self-monitor their blood glucose levels at home. Subsequently, they will input these values directly into a smartphone application called iHealth Gluco-Smart. This application is coupled to a hospital-based platform where these values can be evaluated by the researcher and the endocrinology department.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gestational diabetes mellitus
* Minimum 20 weeks of pregnancy
* Is proficient in Dutch
* Signing the Informed Consent

Exclusion Criteria:

* <20 weeks of pregnancy
* Diagnosis of type 1 diabetes
* Congenital anomalies identified in the fetus
* Participant does not own a smartphone

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Type of delivery (natural or cesarean delivery) in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | After gestation
  Cesarean birth is a maternal risk associated with macrosomia, which is more prevalent in pregnancies complicated with gestational diabetes mellitus. The expected result includes a reduction in cesarean births when incorporating telemonitoring into the standard care of gestational diabetes mellitus compared to the standard care alone.
Number of preterm deliveries in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | After gestation
  Pregnant women with gestational diabetes mellitus are at increased risk of preterm delivery compared to an uncomplicated pregnancy. Proper management of gestational diabetes mellitus could reduce the risk of preterm birth in pregnancies complicated with gestational diabetes mellitus. Therefore, it is expected to have fewer preterm births in the telemonitoring group compared to the control group.
Apgar-score of neonate in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | After gestation
  The Apgar-score serves as an assessment tool for the postnatal health status of newborns. It encompasses five parameters, including: breathing effort, heart rate, muscle tone, grimace response (reflex irritability in response to stimulation), and color. These parameters will be assigned a score on a scale of 0 to 2, where 0 represents a low score and 2 corresponds to the highest score. These scores are then added together to give a total score (maximum 10) that is recorded at 1 minute, and 5 minutes following birth. It is assumed to see higher Apgar-scores in the telemonitoring group compared to the control group, attributable to the enhanced follow-up method.
Birth weight of neonate in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | After gestation
  Macrosomia, defined as a birth weight > 4000 grams, is associated with serious maternal and neonatal adverse outcomes, including cesarean birth and birth fractures, respectively. Therefore, it is important to evaluate the birth weight of neonates. The expected result includes a reduction in birth weight of neonates (< 4000 grams) when incorporating telemonitoring into the standard care of GDM compared to the standard care alone.
Admission to the neonatal intensive care (NIC) in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | After gestation
  Development of gestational diabetes mellitus is associated with neonatal adverse outcomes, including admission tot the neonatal intensive care. The addition of telemonitoring into the standard care process of gestational diabetes mellitus can improve the prenatal follow-up process, potentially impacting neonatal outcomes. It is expected to see fewer admissions to the neonatal intensive care in the telemonitoring group compared to the control group.

SECONDARY OUTCOMES:
Number of prenatal consultations in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | From diagnosis of gestational diabetes mellitus until birth
  Pregnant women with gestational diabetes mellitus are more intensively follow-up compared to an uncomplicated pregnancy. This allows for more efficient monitoring of glycemic values. This in turn enables rapid intervention strategies, such as adjusting diet or increasing insulin units, in response to deviations from desired blood glucose levels. Subsequently, additional prenatal consultations can be reduced in the telemonitoring group compared to the control group.
Number of hospitalizations in pregnancies with gestational diabetes mellitus in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care without telemonitoring. | From diagnosis of gestational diabetes mellitus until birth
  Pregnant women with gestational diabetes mellitus will be hospitalized more often in comparison to an uncomplicated pregnancy. Early detection of gestational diabetes mellitus can make treatment more efficient and reduce the number of hospitalizations. It is expected to see less hospitalizations when adding telemonitoring to the standard care of gestational diabetes mellitus compared to the standard care alone. This reduction can be due to faster response to abnormal blood glucose values and thus less complications.
Reaction time from measuring abnormal glucose values to performing an intervention in pregnancies in which telemonitoring was added to the standard care of gestational diabetes mellitus compared to the standard care alone. | From diagnosis of gestational diabetes mellitus until birth
  The duration between the identification of abnormal glucose values and the implementation of interventions is frequently prolonged due to delayed or absent communication of glucose data. This study will assess whether the addition of telemonitoring in treatment regimens results in a shorter duration for these interventions. Such interventions may encompass dietary adjustments or adjustments to insulin dosages.

OTHER OUTCOMES:
Satisfaction and usability of the modified care process through the administration of patient and staff questionnaires compared to the conventional follow-up approach. | From diagnosis of gestational diabetes mellitus until birth
  Telemonitoring is currently employed in various medical care processes. It aligns more closely with the lifeworld of patients, mitigating the hesitation to make calls and overcoming language barriers. This study will explore potential variations in satisfaction with the monitoring process, aiming to refine and establish an optimal care framework.

CONTACTS AND LOCATIONS:
Overall Officials: Ine Lowyck, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium